CLINICAL TRIAL: NCT05186831
Title: Patient-Portal vs Text-based Hypertension Monitoring Among Black Medicaid/Medicare Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Jennifer Lewey, MD, MPH, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: University of Pennsylvania
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Racial disparities; Digital technology; Hypertension
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text-based monitoring (Experimental): Patients will be asked to take their BP two times daily and text their BP to the study phone number twice a day for 14 days.
  Interventions: Behavioral: Texting
- Online patient portal (Active Comparator): Patients will be asked to take their BP two times daily. They will be given instructions on how to upload BP readings to the online patient portal and will be asked to upload all BP readings. This represents enhanced standard of care.
  Interventions: Behavioral: Online patient portal

INTERVENTIONS:
Behavioral: Texting — Patients will be asked to text their BP. They will receive an automated response to their texts.
  Arms: Text-based monitoring
Behavioral: Online patient portal — Patients will be asked to upload their BP to the online patient portal. They will receive information on how to sign up and use the patient portal. Patients can upload their BP readings daily or at the end of the study period.
  Arms: Online patient portal

SUMMARY:
The coronavirus disease 2019 (COVID-19) pandemic has uprooted conventional health care delivery for routine ambulatory care, requiring health systems to rapidly adopt telemedicine capabilities. The digital divide, has been well documented with lower rates of technology and broadband adoption among racial/ethnic minorities. Additionally, Black patients suffer a disproportionate burden of hypertension and cardiovascular disease. This study will implement a text-based home hypertension monitoring program among Black Medicaid patients with hypertension and cardiovascular disease (CVD) and compare its uptake to the currently available blood pressure monitoring program using the patient portal that is integrated into the electronic health record (EHR).

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Black race
* Medicaid or Medicare insurance
* Hypertension
* Cardiovascular disease or presence of at least 1 cardiovascular risk factor
* Seen for in-person consultation at the Heart and Vascular clinic at the Hospital of the University of Pennsylvania

Exclusion Criteria:

* Does not speak English
* Already owns a BP cuff
* Does not have internet access or a phone 15 with texting capabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Number of BP measurements reported | 14 days
  Number of BP results reported over the study period
Proportion of patients submitting 1 or more BP measurement | 14 days
  Proportion of patients per study arm reporting at least one BP measurement

SECONDARY OUTCOMES:
Patient satisfaction | Within 2 weeks of end of study period
  Patients will be asked to complete a survey about ease of use and likelihood of recommending the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Interested researchers can email study investigator to request de-identified participant data.
Supporting Information: Study Protocol
Time Frame: Study data will be shared within a 4 week timeframe of request.
Access Criteria: Submission of a protocol describing analysis plan.